CLINICAL TRIAL: NCT04284592
Title: Remote Ischemic Postconditioning Increases HIF-1α Plasma Levels and Improves Cardiac Markers After Cardiac Surgery: a Randomised Controlled Study
Brief Title: Remote Ischemic Postconditioning Increases HIF-1α Plasma Levels and Improves Cardiac Markers After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: José García de la Asunción (Other)
Responsible Party: Sponsor-Investigator, José García de la Asunción, Principal investigator and clinical chief, Instituto de Investigacion Sanitaria INCLIVA
Organization: Instituto de Investigacion Sanitaria INCLIVA (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PI07/0836
Record Dates: First submitted 2020-02-21; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Ischemia-reperfusion Injury
Keywords: on-pump cardiac surgery; HIF-1α; Remote ischemic postconditioning; postoperative cardiac markers; cardiopulmonary bypass
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Intervention Model Description: 35 patients receive RIP on upper limb: 5 min of ischemia followed by 5 min of reperfusion (3 cycles) immediately after leaving on-pump. The primary outcome was to know the time course of HIF-1α plasma levels after surgery in both groups and compare the two groups at specific time points: before starting surgery (T0) and after CPB period at 2 h (T1), 8 h (T2), 24 h (T3), 36 h (T4), 48 h (T5). Secondary outcomes included to measure the cardiac markers levels (Troponin T, CK-MB, CPK), arterial oxygenation (PaO2:FiO2) and others.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients do not receive remote ischemic post-conditioning (RIP) after cardiopulmonary bypass
- RIP group (Experimental): Patients receive remote ischemic post-conditioning (RIP) after cardiopulmonary bypass
  Interventions: Procedure: Remote ischemic post-conditioning (RIP)

INTERVENTIONS:
Procedure: Remote ischemic post-conditioning (RIP) — The limb RIP was applied after leaving of cardiopulmonary bypass and consisted of 3 cycles: 5 min of ischemia by a cuff-inflator on an arm and inflated to 200 mmHg, followed by 5 min deflated. The control group had during the same time a deflated cuff.
  Arms: RIP group

SUMMARY:
Background. Cardiopulmonary bypass in on-pump cardiac surgery (OPCS) can have harmful effects by ischemia-reperfusion. No data about the effects of remote ischemic postconditioning (RIP) in hypoxia-inducible factor-1 alpha (HIF-1α) plasma level after OPCS. The aim of this study is evaluate the effects of RIP on postoperative HIF-1α plasma levels, cardiac markers and arterial oxygenation of patients after OPCS.

Methods. Randomised controlled study in 70 patients undergoing OPCS: 35 patients receive RIP (RIP group) and 35 patients not (control group). Patients receive RIP on upper limb: 5 min of ischemia followed by 5 min of reperfusion (3 cycles) immediately after leaving on-pump. The primary outcome was to know the HIF-1α plasma levels after surgery in both groups: before starting surgery (T0) and after CPB period at 2 h (T1), 8 h (T2), 24 h (T3), 36 h (T4), 48 h (T5). Secondary outcomes included to measure the cardiac markers levels (Troponin T, CK-MB, CPK), arterial oxygenation (PaO2/FiO2) and others.

DETAILED DESCRIPTION:
Cardiac surgery with cardiopulmonary bypass (CPB) is associated with ischemia-reperfusion (I-R) injury. Acute myocardial injury after cardiac surgery is associated with increased mortality and morbidity. In 1993, reported that brief circumflex artery occlusion reduces myocardial infarct size induced by a definitive occlusion of the left anterior descending artery, a phenomenon which has been named remote ischemic preconditioning (RIPC). This approach confers resistance to subsequent ischemic episodes in remote organs, possibly by transferring protective mediators through humoral, neuronal, and systemic mechanisms, however the mechanisms involved are not yet fully known. A recent study has found that cardioprotection induced by RIPC the mitochondria appear to be an important subcellular effector organelle. It has been reported that RIPC could be a potential protective approach for perioperative complications. Therefore, the effects on myocardial injury and clinical outcome in patients undergoing on-pump cardiac surgery (OPCS) are inconclusive. In the present study, we conducted a randomized clinical trial on patients undergoing OPCS by application of remote ischemic postconditioning (RIP), an alternative to remote ischemic preconditioning. RIP can be applied in different clinical situations, medical or surgical, when reperfusion is initiated and associated to acidosis, nitric oxide formation, mitochondrial permeability transition pore inhibition and reactive oxygen species generation. In the present study we have opted for remote postconditioning because we speculate a possible losses of plasmatic effectors during CPB procedures using polyvinylchloride (PVC) tubing. Since, when blood is exposed to the PVC surface the plasma proteins may be adsorbed. Also to minimize the bleeding or hemodilution effects on the potential protective plasmatic effectors levels during CPB.

Tissue exposure to low O2 concentration starts a hypoxic response of the hypoxia-inducible factor 1 (HIF-1), a transcription factor heterodimer, consisting of an O2 regulated HIF-1α subunit and a constitutively expressed HIF-1β subunit that binds to the consensus sequence 5'-RCGTG-3', which is present near HIF-1-regulated genes. HIF-1α protein stability is upregulated in response to hypoxia. HIF-1α protein stability is negatively regulated by O2-dependent prolyl hydroxylation and is degraded under normoxia by prolyl hydroxylase. HIF-1α plays a critical role in the mammalian cells activating genes associate with angiogenesis, ischemia, energy metabolism and cell cycle.

The aim of this study carried out in patients undergoing OPCS was the determination of the time course of HIF-1α plasma levels in response to RIP and the possible correlation between aortic cross-clamping time and HIF-1α plasma levels in both groups. HIF-1α role in remote ischemic conditioning (pre or post) is very little known. Therefore, we tested the hypothesis that RIP induces cardiac protection after OPCS and that this is associated to an increase of HIF-1α plasma levels.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery (coronary arteries and/or valve replacement)
* ASA physical status III or less

Exclusion Criteria:

* pregnancy
* previous cardiac surgery
* myocardial infarction (< 6 weeks)
* renal failure
* severe chronic pulmonary disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Study of time course of HIF-1α plasma levels (absorbance units) after on-pump cardiac surgery | Before starting surgery, is the basal time (Time 0)
  Hipoxia induced factor 1 alpha (HIF-1α) is a transcriptional factor. Arterial blood samples were collected from the radial artery to evaluate the changes in HIF-1α plasma levels induced in patients undergoing on-pump cardiac surgery. Because we think that ischemic post-conditioning (RIP) can increase plasma HIF-1α plasma levels.
Study of time course of HIF-1α plasma levels (absorbance units) after on-pump cardiac surgery | 2 hours after cardiopulmonary bypass period (Time 1)
  Hipoxia induced factor 1 alpha (HIF-1α) is a transcriptional factor. Arterial blood samples were collected from the radial artery to evaluate the changes in HIF-1α plasma levels induced in patients undergoing on-pump cardiac surgery. Because we think that ischemic post-conditioning (RIP) can increase plasma HIF-1α plasma levels.
Study of time course of HIF-1α plasma levels (absorbance units) after on-pump cardiac surgery | 8 hours after cardiopulmonary bypass period (Time 2)
  Hipoxia induced factor 1 alpha (HIF-1α) is a transcriptional factor. Arterial blood samples were collected from the radial artery to evaluate the changes in HIF-1α plasma levels induced in patients undergoing on-pump cardiac surgery. Because we think that ischemic post-conditioning (RIP) can increase plasma HIF-1α plasma levels.
Study of time course of HIF-1α plasma levels (absorbance units) after cardiac surgery | 24 hours after cardiopulmonary bypass period (Time 3)
  Hipoxia induced factor 1 alpha (HIF-1α) is a transcriptional factor. Arterial blood samples were collected from the radial artery to evaluate the changes in HIF-1α plasma levels induced in patients undergoing on-pump cardiac surgery. Because we think that ischemic post-conditioning (RIP) can increase plasma HIF-1α plasma levels.
Study of time course of HIF-1α plasma levels (absorbance units) after on-pump cardiac surgery | 36 hours after cardiopulmonary bypass period (Time 4)
  Hipoxia induced factor 1 alpha (HIF-1α) is a transcriptional factor. Arterial blood samples were collected from the radial artery to evaluate the changes in HIF-1α plasma levels induced in patients undergoing on-pump cardiac surgery. Because we think that ischemic post-conditioning (RIP) can increase plasma HIF-1α plasma levels.
Study of time course of HIF-1α plasma levels (absorbance units) after on-pump cardiac surgery | 48 hours after cardiopulmonary bypass period (Time 5).
  Hipoxia induced factor 1 alpha (HIF-1α) is a transcriptional factor. Arterial blood samples were collected from the radial artery to evaluate the changes in HIF-1α plasma levels induced in patients undergoing on-pump cardiac surgery. Because we think that ischemic post-conditioning (RIP) can increase plasma HIF-1α plasma levels.

SECONDARY OUTCOMES:
Study of time course of cardiac marker, Troponin T plasma levels (ng/l) | In summary, not repetitive (6 time points): after anesthetic induction, before starting surgery (Time 0) and after cardiopulmonary bypass period, at 2 hrs (Time 1), 8 hrs (Time 2), 24 hrs (Time 3), 36 hrs (T4), 48 hrs (Time 5).
  Troponin T (ng/l) plasma levels. Similar to HIF-1α measures were studied in six arterial blood samples, which were collected from a radial artery line at 6 specific time points (Time 0 to Time 5).
Study of time course of cardiac marker, creatine phospho-kinase (CPK) plasma levels (U/l) | In summary, not repetitive (6 time points): after anesthetic induction, before starting surgery (Time 0) and after cardiopulmonary bypass period, at 2 hrs (Time 1), 8 hrs (Time 2), 24 hrs (Time 3), 36 hrs (T4), 48 hrs (Time 5).
  Creatine phospho-kinase (CPK) plasma levels (U/l). Similar to HIF-1α measures were studied in six arterial blood samples, which were collected from a radial artery line at 6 specific time points (Time 0 to Time 5).
Study of time course of cardiac marker, creatine kinase-MB (CK-MB) plasma levels (ng/ml) | In summary, not repetitive (6 time points): after anesthetic induction, before starting surgery (Time 0) and after cardiopulmonary bypass period, at 2 hrs (Time 1), 8 hrs (Time 2), 24 hrs (Time 3), 36 hrs (T4), 48 hrs (Time 5).
  Creatine kinase-MB (CK-MB) plasma levels (ng/ml). Similar to HIF-1α measures were studied in six arterial blood samples, which were collected from a radial artery line at 6 specific time points (Time 0 to Time 5).
Study of time course of arterial oxygenation marker (PO2/FiO2), after on-pump cardiac surgery | In summary, not repetitive (6 time points): after anesthetic induction, before starting surgery (Time 0) and after cardiopulmonary bypass period, at 2 hrs (Time 1), 8 hrs (Time 2), 24 hrs (Time 3), 36 hrs (T4), 48 hrs (Time 5).
  Oxygenation marker (PO2/FiO2). Similar to HIF-1α measures were studied in six arterial blood samples, which were collected from a radial artery line at 6 specific time points (Time 0 to Time 5).

CONTACTS AND LOCATIONS:
Overall Officials: José García de la Asunción, MD, PhD, Principal Investigator — Instituto de Investigacion Sanitaria INCLIVA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Przyklenk K, Bauer B, Ovize M, Kloner RA, Whittaker P. Regional ischemic 'preconditioning' protects remote virgin myocardium from subsequent sustained coronary occlusion. Circulation. 1993 Mar;87(3):893-9. doi: 10.1161/01.cir.87.3.893. PMID 7680290
- [Background] Heusch G, Botker HE, Przyklenk K, Redington A, Yellon D. Remote ischemic conditioning. J Am Coll Cardiol. 2015 Jan 20;65(2):177-95. doi: 10.1016/j.jacc.2014.10.031. PMID 25593060
- [Background] Hausenloy DJ, Candilio L, Evans R, Ariti C, Jenkins DP, Kolvekar S, Knight R, Kunst G, Laing C, Nicholas J, Pepper J, Robertson S, Xenou M, Clayton T, Yellon DM; ERICCA Trial Investigators. Remote Ischemic Preconditioning and Outcomes of Cardiac Surgery. N Engl J Med. 2015 Oct 8;373(15):1408-17. doi: 10.1056/NEJMoa1413534. Epub 2015 Oct 5. PMID 26436207
- [Background] Hausenloy DJ, Yellon DM. Ischaemic conditioning and reperfusion injury. Nat Rev Cardiol. 2016 Apr;13(4):193-209. doi: 10.1038/nrcardio.2016.5. Epub 2016 Feb 4. PMID 26843289
- [Background] Wang GL, Jiang BH, Rue EA, Semenza GL. Hypoxia-inducible factor 1 is a basic-helix-loop-helix-PAS heterodimer regulated by cellular O2 tension. Proc Natl Acad Sci U S A. 1995 Jun 6;92(12):5510-4. doi: 10.1073/pnas.92.12.5510. PMID 7539918
- [Background] Garcia-de-la-Asuncion J, Pastor E, Perez-Griera J, Belda FJ, Moreno T, Garcia-del-Olmo E, Marti F. Oxidative stress injury after on-pump cardiac surgery: effects of aortic cross clamp time and type of surgery. Redox Rep. 2013;18(5):193-9. doi: 10.1179/1351000213Y.0000000060. PMID 24020718
- [Background] Kalakech H, Tamareille S, Pons S, Godin-Ribuot D, Carmeliet P, Furber A, Martin V, Berdeaux A, Ghaleh B, Prunier F. Role of hypoxia inducible factor-1alpha in remote limb ischemic preconditioning. J Mol Cell Cardiol. 2013 Dec;65:98-104. doi: 10.1016/j.yjmcc.2013.10.001. Epub 2013 Oct 17. PMID 24140799
- [Background] Cai Z, Luo W, Zhan H, Semenza GL. Hypoxia-inducible factor 1 is required for remote ischemic preconditioning of the heart. Proc Natl Acad Sci U S A. 2013 Oct 22;110(43):17462-7. doi: 10.1073/pnas.1317158110. Epub 2013 Oct 7. PMID 24101519